CLINICAL TRIAL: NCT06134349
Title: The Bipolar Lithium Imaging Scan Study: Imaging Lithium in the Brains of Subjects with Bipolar Disorder
Brief Title: The Bipolar Lithium Imaging Scan Study.
Acronym: BLISS
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: PsyQ (Other); GGZ Rivierduinen (Other)
Responsible Party: Principal Investigator, mleeuw, MD, PhD, Leiden University Medical Center
Other Study IDs: NL80214.058.22
Record Dates: First submitted 2023-11-08; First posted 2023-11-18 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Bipolar Disorder I or II
Keywords: bipolar disorder; lithium; lithium MR imaging; ultra-high field imaging; clinical response; clinical; 7 Tesla
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- BLISS candidates: Adult patients with bipolar disorder (BD) type I or II, who have recently started lithium treatment as part of standard care, will be included. At 12-month follow-up, the longitudinal outcome of lithium treatment will be assessed using a validated questionnaire. Based on previous studies, approximately one-third of participants are expected to be classified as full responders at the 12-month follow-up, with another one-third classified as clinical non-responders to lithium treatment.
  Interventions: Other: Lithium MR imaging

INTERVENTIONS:
Other: Lithium MR imaging — After obtaining written informed consent and within four weeks of reaching a stable therapeutic serum lithium concentration, lithium MR imaging will be performed using a 7 Tesla MR system (Achieva, Philips Medical Systems, Eindhoven, The Netherlands) with a dual-tuned 7Li/1H volume head coil (RAPID Biomedical GmbH, Rimpar, Germany). Various approaches, including whole-brain, voxel-wise, parcellation, mean, and regions of interest, will be applied to measure lithium concentrations.

SUMMARY:
The main goal of this study is to determine if brain lithium-concentrations predict clinical lithium treatment-response. Secondary, to study correlations between intracerebral distribution-patterns of lithium with clinical treatment outcome.

Brain lithium concentrations will be measured using ultra-high field (7 Tesla) lithium magnetic resonance (MR) imaging, which has recently been introduced. Determining lithium-concentrations in the brain has been difficult so far due to lithium's relatively low concentration (compared to protons, which are targeted in conventional MRI). 7T lithium MR imaging has the potential to produce much more detailed MR images compared with previous studies, for the first time. The BLISS study is expected to yield new insights, helping to better understand why clinical lithium response varies between individuals.

DETAILED DESCRIPTION:
Introduction Lithium treatment is considered the first-line pharmacological treatment for bipolar disorder. However, individual responses vary greatly, which undermines the ability to achieve rapid stabilization in many patients with bipolar disorder. The neurobiological mechanisms underlying lithium's action are still largely unknown, which hampers the development of clinically applicable predictors for individual treatment response. The recent introduction of ultra-high-field lithium magnetic resonance imaging offers a promising avenue to better link brain measures with clinical responses to lithium treatment.

Methods and Analysis This is a longitudinal observational study involving 80 adults with bipolar disorder who are initiating lithium as part of their regular treatment regimen. Ultra-high-field lithium magnetic resonance imaging of the brain will be performed within four weeks of reaching stable therapeutic serum lithium concentrations. The primary outcome is clinical response to lithium treatment at one-year follow-up, as measured using a validated questionnaire. Linear regression analysis will be used to establish correlations between brain lithium concentrations-including whole brain, voxel-wise, parcellation, mean, and region-of-interest approaches-and clinical lithium response.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 years or above,
2. a clinical diagnosis of bipolar disorder type I or type II ,
3. having reached stable therapeutic serum lithium concentrations (reference values 0.6-1.0 mM in age to 65 years; 0.4-0.8 in age 65 years and above) within four weeks prior to study participation, and
4. provided written informed consent.

Exclusion Criteria:

1. insufficient comprehension of the Dutch language,
2. unable to provide informed consent,
3. drug or alcohol abuse over a period of two weeks prior to study participation, and
4. meeting any exclusion criterium for MR imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with bipolar disorder type I or II who start with lithium treatment as part of standard care.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Clinical lithium response | At 12-month follow-up.
  Clinical lithium response will be assessed using a validated questionnaire.

SECONDARY OUTCOMES:
Serum lithium concentrations | Baseline
  Serum lithium concentrations will be determined to establish correlations with brain lithium concentrations.

OTHER OUTCOMES:
Manic and depressive symptom severity | Baseline
  Manic and depressive symptom rating scales will be used to assess mood state at the day of scan acquisition.

CONTACTS AND LOCATIONS:
Overall Officials: E Boere, MD, Study Chair — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Lithium MR imaging data.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: Study protocol - currently submitted for OA publication CSR - after termination of the BLISS study Analytic code - after termination of the BLISS study IPD - after termination of the BLISS study
Access Criteria: Study protocol - open access CSR and analytic code - open access
  IPD: lithium imaging data will be made available upon request with the study chair, and no sooner then after study termination.

REFERENCES:
- [Derived] Boere E, van der Wee NJA, van Hemert AM, Webb AG, de Leeuw M. The Bipolar Lithium Imaging Scan Study (BLISS): protocol for a 7T lithium-7 magnetic resonance study in bipolar disorder. Psychoradiology. 2025 Mar 7;5:kkaf003. doi: 10.1093/psyrad/kkaf003. eCollection 2025. PMID 40160802